CLINICAL TRIAL: NCT03766295
Title: A Prospective, Multicenter, Double-randomized, Double-blind, 2-parallel Groups, Phase 3 Study to Compare as First Line Therapy Efficacy and Safety of Masitinib in Combination With Gemcitabine, to Gemcitabine in Combination With Placebo, in the Treatment of Patients With Non Resectable Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Masitinib Plus Gemcitabine in Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB12005
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Locally Advanced or Metastatic Pancreatic Cancer
Keywords: Pancreatic cancer; tyrosine kinase inhibitor
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — masitinib; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- Masitinib & gemcitabine (Experimental): Participants receive masitinib (6 mg/kg/day), given orally twice daily, plus gemcitabine at 1000mg/m2 by intravenous infusion during 30 minutes, once every 7 days, for up to 7 weeks, followed by a week of rest. Subsequent cycles should consist of an IV infusion, once every 7 days, for 3 consecutive weeks out of every 4 weeks, until disease progression, death, limiting toxicity or patient consent withdrawal.
  Interventions: Drug: Masitinib; Drug: Gemcitabine
- Placebo & gemcitabine (Active Comparator): Participants receive matching placebo, given orally twice daily, plus gemcitabine at 1000mg/m2 by intravenous infusion during 30 minutes, once every 7 days, for up to 7 weeks, followed by a week of rest. Subsequent cycles should consist of an IV infusion, once every 7 days, for 3 consecutive weeks out of every 4 weeks, until disease progression, death, limiting toxicity or patient consent withdrawal.
  Interventions: Drug: Gemcitabine; Drug: Placebo

INTERVENTIONS:
Drug: Masitinib
  Other Names: AB1010
  Arms: Masitinib & gemcitabine
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Placebo
  Other Names: Placebo Oral Tablet
  Arms: Placebo & gemcitabine

SUMMARY:
The objective is to compare efficacy and safety of masitinib in combination with gemcitabine to placebo in combination with gemcitabine, in treatment of patients with locally advanced or metastatic pancreatic cancer and who have pain related to the disease.

DETAILED DESCRIPTION:
Masitinib is a selective tyrosine kinase inhibitor that is thought to promote survival via modulation of immunostimulation-mediated anticancer effects and modulation of the tumor microenvironment. The objective of this study is to evaluate the efficacy and safety of masitinib in combination with gemcitabine with respect to placebo in combination with gemcitabine for the treatment of non resectable locally advanced or metastatic pancreatic cancer patients with pain related to the disease. Approximately 330 patients with pain Visual Analogue Scale (VAS) > 20 and/or treated with 'opioid analgesics' dose ≥ 1 mg/kg/day at baseline will be randomized in a 2:1 ratio to the masitinib and placebo arms, respectively. The primary outcome measure is overall survival (OS).

ELIGIBILITY:
Main inclusion criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the pancreas, non resectable locally advanced or metastatic stage
2. Patient with pain related to the disease, as assessed by the investigator and the patient:

   * Pain related to the disease as assessed by the investigator is defined as clinical and documented evaluation by the investigator during physical examinations at screening and/or baseline.
   * Pain, as assessed by the patient is defined as at least one value out of two values > 20mm on Visual Analogue Scale at screening or baseline. Visual Analogic scale consists in the visual representation of pain amplitude as perceived by the patient. The amplitude is represented by a 100 mm long line having no reference marks. One extremity indicates an absence of pain (0 value) and the other the worst imaginable pain (100 value).

OR

- Patient treated with opioid analgesics at a dose ≥ 1 mg/kg/day (morphinic equivalent).

3. Chemotherapy naïve patient for the advanced/metastatic disease

Main exclusion criteria:

1. Patient with no pain related to the disease (as defined in the inclusion criterion number 2)
2. Pregnant or nursing female patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival (median) | From day of randomization to death, assessed for a maximum of 60 months
  Overall survival is defined as time in months from the randomization date to the date of death due to any cause. If a patient is not known to have died, then OS will be censored at the date of last known date patient alive.

SECONDARY OUTCOMES:
Survival rates | every 24 weeks
  The proportion of patients alive at each time point, estimated with Kaplan-Meier distribution
Progression Free Survival | From day of randomization to disease progression or death, assessed for a maximum of 60 months
  Progression Free Survival (PFS) is defined as the time from the randomization date until the date of earliest evidence of disease progression or death, for participants who progressed or died before subsequent cancer therapy. Disease progression will be assessed by the investigator on CT scan according to RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Joël Ezenfis, MD, Principal Investigator — Centre Hospitalier de Longjumeau, France
Locations (9):
- Hospital AZ Sint-Jan, Bruges, Belgium
- France (2):
  - Polyclinique de Limoges site CHENIEUX, Limoges
  - Centre Hospitalier de Longjumeau, Longjumeau
- General University Hospital of Patras, Pátrai, Greece
- Sanjeevani CBCC USA Cancer Hospital, Raipur, India
- Omsk Clinical oncology dispensary Omsk, Omsk, Russia
- National Oncology Institute, Bratislava, Slovakia
- Institut Salah Azaiez de Cancerologie, Bab Saadoun, Tunisia
- Center of Surgical Innovations, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided